CLINICAL TRIAL: NCT02792283
Title: Evaluation of the Bleeding Risk in Patient Undergoing Hemodialysis by the Analysis of Platelet Function by PFA-100®
Brief Title: Platelet Function in Hemodialysis Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PA15098
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

ARMS (1):
- patients undergoing hemodialysis (Experimental)
  Interventions: Biological: whole blood collection

INTERVENTIONS:
Biological: whole blood collection

SUMMARY:
The objective is to evaluate the function of the platelet in patients undergoing hemodialysis. The investigators will use the assay called PFA-100, an in vitro whole blood assay with three pathways of platelet activation to describe a platelet response profile.

The hypothesis is that patients undergoing hemodialysis present a platelet dysfunction, that may be reversed by hemodialysis. The effect of heparin, used during hemodialysis session to anticoagulate the hemodialyzer, on platelet function will be assessed.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the platelet function during hemodialysis. One hundred patients with end-stage renal disease undergoing hemodialysis (2 to 3 sessions per week, 3 to 4 hours per session) will be included.

Patients who meet the inclusion criteria will be included after oral and written information and signature of written consent.

The study consists in recording clinical and biological and the evaluation of platelet function by the PFA-100 assay. This is a whole blood platelet function assay, with 3 pathways of platelet activation (collagen-epinephrine, collagen-ADP and specific P2Y cartridge - Innovance®).

Whole blood is collected in the arterial line of the arteriovenous vascular access (fistula or graft) before and after the hemodialysis session.

PFA-100 is assayed within 2 hours after blood collection and the platelet response profile is interpreted according to the manufacturers instructions.

Clinical informations, especially hemorragic and thrombotic history, are collected the day of inclusion and 6 months after inclusion.

ELIGIBILITY:
Inclusion criteria :

patient with end-stage chronic kidney disease undergoing hemodialysis age ≥ 18 years old hemodialysis on a peripheral vascular access (arteriovenous fistula or graft) hematocrit between 0.35 and 0.50 and platelet count between 150 and 500 G/L written consent after oral and written information

Exclusion criteria :

pregnancy, breast feeding legal guardianchip hemodialysis on a catheter inability to sign the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
PFA-100 quantification | at the day of inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France